CLINICAL TRIAL: NCT04294212
Title: Medical Termination of Pregnancy : Evaluation of Patients' Practices and Feelings in Brest Hospital
Acronym: IMGEPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMGEPR (29BRC19.0245)
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-03

CONDITIONS: Medical Termination of Pregnancy
Keywords: Pregnancy loss; lived from patients; medical termination of pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate the feelings of patients about a medical termination of pregnancy that they experienced in Brest Hospital. Patients responded to an online questionnaire assessing their feelings at each stage of the medical termination process. Their answers were associated with their medical data.

ELIGIBILITY:
Inclusion Criteria:

* Patient having experienced a medical termination of pregnancy in Brest Hospital
* Medical termination of pregnancy after 14 weeks
* Induction for natural delivery
* No opposition

Exclusion Criteria:

* Medical termination of pregnancy before 14 weeks
* Selective termination of pregnancy (multiple pregnancy)
* Caesarean
* Patient not speaking french
* Patient's refusal

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients having experienced a medical termination of pregnancy in Brest Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall satisfaction score | One day
  answers to a satisfaction questionnaire based on a numerical scale ranging from 0 (dissatisfaction) to 3 (satisfaction), then calculation of the overall score

SECONDARY OUTCOMES:
satisfaction score by indicator | One day
  satisfaction questionnaire divided into several parts according to an indicator

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement